CLINICAL TRIAL: NCT03810859
Title: Non-syndromic Inherited Anomalies of Mineralized Tooth Tissues: a Whole Exome Study to Identify New Pathogenic Variants
Acronym: EXODENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French rare diseases Healthcare Network (Unknown); The French Foundation for Rare Diseases (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: K180404J; 2018-A01250-55 (Other: ID-RCB)
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Amelogenesis Imperfecta; Dentinogenesis Imperfecta; Dentin Anomalies
Keywords: Amelogenesis imperfecta; Dentinogenesis imperfecta; Dentin anomalies; Whole Exome Study
MeSH Terms: conditions — Amelogenesis Imperfecta; Dentinogenesis Imperfecta | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): Blood sample
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Adults : 7 to 10 mL Childs : 2 to 4 mL

SUMMARY:
ExoDent specifically aims to discover new genes and new mutations causing isolated amelogenesis imperfecta (AI) and dentinogenesis imperfecta (DI) and other dentin anomalies. The key point for clinicians is to distinguish between non syndromic and syndromic disorders in order to improve patients guidance and counseling. To do so, two targeted NGS panel have been designed, one searching for isolated AI and the other for DI. After 18 months, some families remain without any positive results. ExoDent project proposes those negative patients a Whole Exome Sequencing (WES) approach to deeper explore their genetic background.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of amelogenesis imperfecta or dentinogenesis imerfecta or other dentin anomaly with no other signs or symptoms ( familial or isolated)
* negative results after targeted NGS strategy for molecular diagnosis

Exclusion Criteria:

* absence of positive clinical diagnosis
* Diagnosis of syndromic disease

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Genome sequencing | After one day
  Pathogenic variants identification and qualification

CONTACTS AND LOCATIONS:
Overall Officials: Céline GAUCHER, MD, Principal Investigator — APHP
Locations (1):
- Hospital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No